CLINICAL TRIAL: NCT07083466
Title: Assessment of Composite Inflammatory Ratios in Juvenile Idiopathic Arthritis and Their Association With Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hadeer Fadlalmawla Mohamed, resident at rheumatology and rehabilitation department at sohag university hospitals, Sohag University
Other Study IDs: Soh-Med-25-6-6MS
Record Dates: First submitted 2025-06-27; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- case: cases under 16y established diagnosis juvenile idiopathic arthritis
  Interventions: Diagnostic Test: complete blood count; Diagnostic Test: serum albumin
- control: below age 16 y not diagnosed with any autoimmune or systemic disease
  Interventions: Diagnostic Test: complete blood count; Diagnostic Test: serum albumin

INTERVENTIONS:
Diagnostic Test: complete blood count — blood test
Diagnostic Test: serum albumin — blood test

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is a prevalent pediatric rheumatic disorder characterized by persistent inflammation of one or more joints in children and adolescents. This chronic condition is a major contributor to both short- and long-term morbidity and functional disability We aim in this study to investigate the role of CAR, PLR, NLR ,systemic inflammatory index (SII ) and NAR ( SII and NAR have never been evaluated before in JIA patients ) as potential markers of disease activity in patients with non-systemic JIA (nsJIA) .

ELIGIBILITY:
Inclusion Criteria:

-

1. Patients who classified JIA according to International League of Associations for Rheumatology ILAR criteria on treatment with exclusion of systemic JIA.

2. Patients with disease duration more than 6 months. 3. Age below 16 years old. 4. Patient cooperative and can answer questions. 5. Patients who are able and willing to give written informed consent or their parents/guardians

Exclusion Criteria:

* 1. Systemic JIA. 2. Patients with other autoimmune or autoinflammatory diseases, immunodeficiencies, hematologic conditions, malignances and infectious disease at enrollment time or in the previous 2 weeks.

Patients who are not able and willing to give written informed consent

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include 60 patients classified as JIA according International League of Associations for Rheumatology ILAR criteria on treatment who will recruited from Rheumatology and Rehabilitation department at Sohag University hospital in addition to 30 healthy individual volunteers without history of any systemic active disease recruited from the community as age and sex matched controls
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
possibility to use crp to albumin level as novel biomarker to predict disease activity in juvenile 0idiopathic arthritis | 6 months
possibility to detect systemic inflammatory index and its relation to disease activity and risk of flare in juvenile idiopathic arthritis | 6 months
assessment of activity of disease according to JDAS SCORE | 6 months
assessment of neutrophils to albumin ratio and its relation to JDAS score activity score | 6 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang JL. New advances in juvenile idiopathic arthritis. Chang Gung Med J. 2012 Jan-Feb;35(1):1-14. doi: 10.4103/2319-4170.106171. PMID 22483423
- [Background] Prakken B, Albani S, Martini A. Juvenile idiopathic arthritis. Lancet. 2011 Jun 18;377(9783):2138-49. doi: 10.1016/S0140-6736(11)60244-4. PMID 21684384
- [Background] Milovanovic M, Nilsson E, Jaremo P. Relationships between platelets and inflammatory markers in rheumatoid arthritis. Clin Chim Acta. 2004 May;343(1-2):237-40. doi: 10.1016/j.cccn.2003.12.030. PMID 15115702
- [Background] Erre GL, Paliogiannis P, Castagna F, Mangoni AA, Carru C, Passiu G, Zinellu A. Meta-analysis of neutrophil-to-lymphocyte and platelet-to-lymphocyte ratio in rheumatoid arthritis. Eur J Clin Invest. 2019 Jan;49(1):e13037. doi: 10.1111/eci.13037. Epub 2018 Nov 6. PMID 30316204